CLINICAL TRIAL: NCT06605989
Title: The Effect of Nostril Side on Epistaxis During Nasotracheal Intubation
Brief Title: Nostril Side on Epistaxis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-2024-0025
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-09

CONDITIONS: Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- left nostril side (Experimental): For nasotracheal intubation, the nasal RAE tube will be inserted through the left nostril and advanced into the oral cavity.
  Interventions: Procedure: Nasotracheal intubation
- right nostril side (Experimental): For nasotracheal intubation, the nasal RAE tube will be inserted through the right nostril and advanced into the oral cavity.
  Interventions: Procedure: Nasotracheal intubation

INTERVENTIONS:
Procedure: Nasotracheal intubation — For nasotracheal intubation, the nasal RAE tube will be first inserted through the left nostril for patients in the left nostril side arm. For nasotracheal intubation, the nasal RAE tube will be first inserted through the right nostril for patients in the right nostril side arm.

SUMMARY:
The purpose of the study is to investigate the effect of the nostril side on epistaxis during nasotracheal intubation.

DETAILED DESCRIPTION:
This prospective randomized controlled study was approved by the IRB of our institute.

Patients requiring nasotracheal intubation will be screened for eligibility for the study. Then, patients will be randomized to one of two groups; (Group I: tube will be inserted through the left nostril and advanced into the oral cavity / Group II: tube will be inserted through the right nostril and advanced into the oral cavity). After induction of anesthesia and muscle relaxation, the preformed nasal RAE (Ring-Adair-Elwyn) tube will be inserted via the nostril, which is assigned to each patient according to the group, approximately 3-4 cm. Next, an anesthesiologist will advance the tube into the oral cavity. After the tube is placed in the oral cavity, the anesthesiologist will perform nasotracheal intubation with Magill forceps. After that, an investigator will check the occurrence of epistaxis due to nasotracheal intubation and its severity with a fiberoptic bronchoscope. After obtaining all data, investigators will analyze the incidence of epistaxis and its severity between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients requiring nasotracheal intubation for elective surgery

Exclusion Criteria:

* refuse to participate in the study
* severe deformity in the nose
* current severe epistaxis
* cannot insert the tube into a specific nostril side due to any reason

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
epistaxis | during nasotracheal intubation
  epistaxis due to nasotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,Ph.D., Principal Investigator — Seoul National University College of Medicine, Seoul Metropolitan Government Seoul National University Boramae Medical Center
Locations (2):
- South Korea (2):
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Dongjak-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sanuki T, Hirokane M, Kotani J. Epistaxis during nasotracheal intubation: a comparison of nostril sides. J Oral Maxillofac Surg. 2010 Mar;68(3):618-21. doi: 10.1016/j.joms.2009.04.097. Epub 2009 Nov 22. PMID 19931965